CLINICAL TRIAL: NCT04696952
Title: A Driving Performance Evaluation Study of TS-142 Using a Driving Simulator in Non-elderly and Elderly Healthy Subjects
Brief Title: A Study to Evaluate Next Day Effects of TS-142 on Driving Performance in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TS142-207
Record Dates: First submitted 2020-12-18; First posted 2021-01-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — TS-142; zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TS-142 10 mg (Experimental): Period in which subjects received TS-142 10 mg
  Interventions: Drug: TS-142
- TS-142 20 mg (Experimental): Period in which subjects received TS-142 20 mg
  Interventions: Drug: TS-142
- Zopiclone 7.5 mg (Experimental): Period in which subjects received Zopiclone 7.5 mg
  Interventions: Drug: Zopiclone
- Placebo (Experimental): Period in which subjects received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-142 — TS-142
  Arms: TS-142 10 mg; TS-142 20 mg
Drug: Zopiclone — Zopiclone
  Arms: Zopiclone 7.5 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A clinical study to evaluate the residual effects of TS-142 on driving performance in healthy and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 21 years or older but less than 80 years at the time of informed consent
* Those with a BMI of 18.5 or more and less than 25.0 and a body weight of 40.0 kg or more at screening tests
* Have an ordinary driving license and have driven on a daily basis for more than 3 years
* Have a constant sleep pattern (waking up from 5:00 to 9:00, falling asleep from 21:00 to 1:00 and time in bed is from 6 to 8 hours)
* No visual impairment (those who have >=0.7 vision in both eyes and >=0.3 in each eye at vision test of screening tests, enable to correct the vision with eyeglasses or contact lens)
* Those who have cognitive and physical function (adequate dexterity of fingers, vision and hearing etc.) to operate Driving Simulator (DS) certainly, understand and carry out the direction on the task of the DS evaluation
* Those with no abnormal findings in medical examinations, vital signs, or 12-lead electrocardiogram and whose laboratory test results were within the reference values of the study site based on the results of screening tests and tests obtained before hospitalization of Visit 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Those who have any disease and are not regarded as healthy subjects based on the medical judgment of the principal investigator or sub-investigator
* Those who have a medical history that makes them ineligible for participation in this study such as respiratory disease, cardiovascular disease, gastrointestinal disease, liver disorder, renal disorder, urological disease, endocrine disease, metabolic disease, hematological disease, immune disease, skin disease, neurological disease, mental disorder etc.
* Those who have had symptoms of parasomnia (parasomnia, sleepwalking, abnormal dreams, nightmares), narcolepsy-like symptoms (cataplexy, hypnagogic hallucinations, sleep paralysis), or suicide attempt
* Those who have hypersensitivity to zopiclone or s-zopiclone
* Those who have experienced a time difference of 6 hours or more within 1 week prior to Visit 1, or who will be exposed to such time difference during the study period
* Those who have performed irregular shift work or night shift work within 4 weeks prior to Visit 1, or need to do so during the study period
* Those who have performed the DS evaluation used in this clinical trial in the past
* Those who received TS-142 (active drug) in the past
* Those who go of course even once at the DS evaluation in Visit1
* Those whose total SDLP in 60 minutes at the DS evaluation in Visit1 is more than 60 cm
* Other protocol defined exclusion criteria could apply

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Standard deviation of lateral position (SDLP) evaluated by using a driving simulator on day 2 | On day 2 at 9 hours post dose
Standard deviation of lateral position (SDLP) evaluated by using a driving simulator on day 9 | On day 9 at 9 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No